CLINICAL TRIAL: NCT01780896
Title: The Relationship Between Vestibular Function and Topographic Memory
Brief Title: Relationship Between Vestibular Function and Topographic Memory
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Michael Roman, PhD, LSSD (Unknown); Ears of Texas, PA (Unknown)
Responsible Party: Sponsor
Other Study IDs: 121101-R43TR000645-01; R43TR000645 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Normal Elderly Population
Keywords: Topographical Memory; Non-Topographical Memory; Vestibular Function; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group

SUMMARY:
The purpose of this study is to evaluate visual and nonvisual topographic memory impairment and its relationship to vestibular function in humans. Topographic memory refers to the ability to remember current and past locations in topographic (navigational) space and to make and/or adjust to spatial transformations using such memories. Performance on each of these topographic memory tasks will be compared to performance on a set of comparable nontopographic memory tasks. Topographic impairments represent some of the earliest cognitive deficits observed in Alzheimer's Disease, and the brain areas involved in topographic memory are the first to show degenerative changes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of all racial and ethnic groups between the ages of 70 and 85 years of age;
* Montreal Cognitive Assessment (MOCA) (http://www.mocatest.org) score of >24;
* No known history or current evidence of stroke, trauma, psychiatric illness, or other insult to the brain;
* No current use of psychoactive medicine other than caffeine (100 mg/day) or alcohol (1-2 drinks per night);
* Normal sleep (at least an average of 7 hours for four days prior to participation);
* Able and willing to comply with study requirements including following instructions to complete vestibular and neuropsychological testing; and
* Have full understanding of all elements of provide signature and dating of the written informed consent prior to the initiation of procedures specified in protocol.

Exclusion Criteria:

* <70 or >85 yrs of age;
* MOCA score of <25;
* History, or current evidence, of stroke, trauma, psychiatric illness, or other insult to the brain;
* Prior history of inner-ear balance problems;
* Current use of psychoactive medicine other than moderate caffeine or alcohol use;
* Acute or chronic sleep deprivation during the week prior to participation (<7 hours/night on average for four nights prior to participation).

Other Restrictions:

* No alcohol use on the night before the vestibular testing
* 7 hours minimum sleep the night before vestibular testing
* No eye make-up can be worn on the day of the vestibular test due to possible interference with vestibular-ocular reflex testing apparatus

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Nominally healthy adults between the ages of 70 and 85 yrs who meet inclusion/exclusion criteria. All study participants will be recruited from the San Antonio community.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Determine relationship between topographic memory and vestibular function | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Fred Previc, PhD, Principal Investigator — Biomedical Development Corporation
Locations (2):
- United States (2):
  - Ears of Texas, PA, San Antonio, Texas
  - Michael Roman, PhD, LSSP, San Antonio, Texas